CLINICAL TRIAL: NCT04400344
Title: Approaches to Foot Complication Prevention: A Survey of Diabetes Educators
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Podimetrics, Inc. (Industry)
Collaborators: American Association of Diabetes Educators (Other)
Responsible Party: Sponsor
Other Study IDs: A20-018-682
Record Dates: First submitted 2020-05-18; First posted 2020-05-22 (Actual); Last update posted 2020-08-31 (Actual); Status verified 2020-08

CONDITIONS: Foot Ulcer, Diabetic
Keywords: Diabetic Foot; Ulcer; Care recommendation; Foot Diseases; Diabetic Neuropathies; Diabetes Education; Diabetes; Diabetes Educator; Diabetes Mellitus; Diabetes Complication; Care and treatment
MeSH Terms: conditions — Diabetic Foot; Ulcer; Foot Diseases; Diabetic Neuropathies; Diabetes Mellitus; Diabetes Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Survey Respondents: Respondents are members of the American Association of Diabetes Educators recruited via an introductory email sent out by the AADE on behalf of Podimetrics.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The purpose of the survey is to assess the knowledge base, role in management, and resources available to diabetes educators regarding foot complication prevention within a variety of healthcare settings.

DETAILED DESCRIPTION:
Podimetrics is a care management company with a temperature-based foot monitoring solution to help prevent diabetic foot ulcers, one of the most debilitating and costly complications of diabetes.

Diabetes educators within the AADE/ADCES encompass a wide array of medical disciplines including nurses, physicians, dieticians, and pharmacists. Diabetes researchers want to better understand the degree to which diabetic foot care and prevention is incorporated into the diabetes education curriculum. To what extent are these topics discussed between diabetes educators and the patients they interact with? And how comfortable are educators in discussing these topics?

To gain insight into these questions Podimetrics researchers have designed an online questionnaire survey for completion by AADE members. The general purpose of the survey is to assess the knowledge base, role in management, and resources available to diabetes educators regarding foot complication prevention within a variety of healthcare settings.

The specific aim is to collect generalizable data to characterize the current state of diabetic foot education and identify any gaps in knowledge that may be present. Furthermore, if it is found that educators are lacking important knowledge which supports ample diabetic foot health education, approaches to bridge these gaps may be suggested through published recommendations.

ELIGIBILITY:
Inclusion Criteria:

* American Association of Diabetes Educators (AADE) member with accurate email address on file with the AADE.

Exclusion Criteria:

* AADE member with an inability to read English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Respondents are members of the American Association of Diabetes Educators (AADE) recruited via an introductory email sent out by the AADE on behalf of Podimetrics.
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2020-06-13 (Actual); Primary Completion 2021-05-13 (Estimated); Study Completion 2021-05-13 (Estimated)

PRIMARY OUTCOMES:
Current state of diabetic foot care education and knowledge base among diabetic educators | One year
  Survey of diabetic foot care recommendations, treatment options, risk classifications, role in management, and resources available to diabetes educators regarding foot complication prevention within a variety of healthcare settings.

CONTACTS AND LOCATIONS:
Locations (1):
- Podimetrics,Inc., Somerville, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
To protect the respondent's identity, respondent name and email address will not be recorded within the survey results. No demographic data other than relevant profession, work environment, and number of years as a certified educator will be collected. Additionally, the AADE will not share respondent's name or email addresses with Podimetrics, and the AADE will not have access to the individual survey results, effectively detaching individual results from respondents' identities.